CLINICAL TRIAL: NCT00128388
Title: Randomized Controlled Trial of Psychodynamic Psychotherapy vs. Applied Relaxation for Panic Disorder
Brief Title: Psychodynamic Therapy for Treating Panic Disorder
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Barbara Milrod, M.D., Professor of Psychiatry, Weill Medical College of Cornell University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K23MH001849 (NIH); K23MH001849 (NIH); DSIR AT-CD
Record Dates: First submitted 2005-08-05; First posted 2005-08-09 (Estimated); Last update posted 2013-06-27 (Estimated); Status verified 2013-06

CONDITIONS: Panic Disorder
Keywords: panic disorder,; psychodynamic psychotherapy,; efficacy trial
MeSH Terms: conditions — Panic Disorder | interventions — Psychotherapy, Psychodynamic; Behavior Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 PFPP (Experimental): Panic Focused Psychodynamic Psychotherapy
  Interventions: Other: PFPP
- 2 ART (Active Comparator): Applied Relaxation Training
  Interventions: Other: ART

INTERVENTIONS:
Other: PFPP — Psychoanalytic Psychotherapy for panic disorder
  Other Names: Psychodynamic psychotherapy
  Arms: 1 PFPP
Other: ART — Applied Relaxation Training
  Other Names: Applied Relaxation Training; Behavioral Therapy
  Arms: 2 ART

SUMMARY:
This study will determine the effectiveness of a manualized form of brief psychodynamic psychotherapy in comparison with applied relaxation training in treating adults with panic disorder.

DETAILED DESCRIPTION:
This is a randomized controlled trial of a manualized form of brief psychodynamic psychotherapy in comparison with applied relaxation training, a less active form of treatment in other studies, for adults with primary Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) panic disorder.

Forty nine patients who have signed written consent who have primary DSM-IV panic disorder have been entered into the study. Randomization has been stratified by presence of major depression and use of psychoactive, anti-panic medications. Medications, if present, have been held constant. All patients have received 24 sessions of either psychodynamic psychotherapy, or applied relaxation training for panic disorder. This study is currently closed for recruitment, although final follow-up assessments have yet to be completed.

ELIGIBILITY:
Inclusion Criteria:

* 18-55 years old
* Primary DSM-IV panic disorder with or without agoraphobia
* Severity 5/8 minimum on the Anxiety Disorders Interview Schedule

Exclusion Criteria:

* Psychosis
* Unstable medication dosage
* Unwilling to discontinue ongoing psychotherapy
* Organic mental syndrome
* Substance use or abuse

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2000-02; Primary Completion 2005-01 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
PDSS (panic disorder severity scale) | termination, 2, 4, 6, 12 month f/u

SECONDARY OUTCOMES:
SDS (Sheehan disability scale) | termination, 2, 4, 6, 12 month f/u
HARS (Hamilton anxiety rating scale) | termination, 2, 4, 6, 12 month f/u
HDRS (Hamilton depression rating scale) | termination, 2, 4, 6, 12 month f/u

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Milrod, M.D., Principal Investigator — Weill Medical College
Locations (1):
- Weill Medical College, New York, New York, United States

REFERENCES:
- [Derived] Gibbon S, Khalifa NR, Cheung NH, Vollm BA, McCarthy L. Psychological interventions for antisocial personality disorder. Cochrane Database Syst Rev. 2020 Sep 3;9(9):CD007668. doi: 10.1002/14651858.CD007668.pub3. PMID 32880104
- [Derived] Klass ET, Milrod BL, Leon AC, Kay SJ, Schwalberg M, Li C, Markowitz JC. Does interpersonal loss preceding panic disorder onset moderate response to psychotherapy? An exploratory study. J Clin Psychiatry. 2009 Mar;70(3):406-11. doi: 10.4088/jcp.08m04248. Epub 2008 Nov 18. PMID 19026262
- [Derived] Milrod BL, Leon AC, Barber JP, Markowitz JC, Graf E. Do comorbid personality disorders moderate panic-focused psychotherapy? An exploratory examination of the American Psychiatric Association practice guideline. J Clin Psychiatry. 2007 Jun;68(6):885-91. doi: 10.4088/jcp.v68n0610. PMID 17592913